CLINICAL TRIAL: NCT06702111
Title: Allogeneic Hematopoietic Stem Cell Transplant (HSCT) in Adults: Clinical Outcome and Complications
Brief Title: Outcome of Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: ALLO-HSCT-001
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hematopoietic Stem Cell Transplant (HSCT)
Keywords: Hematopoietic stem cell transplantation; Prognostic factors; Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients receiving allogeneic HSCT at Queen Mary Hospital, Hong Kong

SUMMARY:
To collect baseline and outcome data relating to all bone marrow, peripheral blood, cord blood hematopoietic stem cell transplants and therapies related to hematopoietic stem cell transplantation performed in Queen Mary Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older who received allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Exclusion Criteria:

* participant who is unable to give informed consent in a prospective cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years or older who are undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT) at Queen Mary Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 year
  Time from HSCT to death or latest follow-up
Relapse-free survival | 5 years
  Time from HSCT to relapse, death or latest follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Harry HS Gill, MBBS, MD, FRCP, FRCPath, Principal Investigator — Department of Medicine, the University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Medicine, Queen Mary Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared based on institutional policies.

REFERENCES:
- [Background] Passweg JR, Baldomero H, Chabannon C, Basak GW, de la Camara R, Corbacioglu S, Dolstra H, Duarte R, Glass B, Greco R, Lankester AC, Mohty M, Peffault de Latour R, Snowden JA, Yakoub-Agha I, Kroger N; European Society for Blood and Marrow Transplantation (EBMT). Hematopoietic cell transplantation and cellular therapy survey of the EBMT: monitoring of activities and trends over 30 years. Bone Marrow Transplant. 2021 Jul;56(7):1651-1664. doi: 10.1038/s41409-021-01227-8. Epub 2021 Feb 23. PMID 33623153